CLINICAL TRIAL: NCT01667796
Title: Pharmacodynamic and Immunologic Effects of Vitamin D Supplementation in Patients With Multiple Sclerosis and Healthy Controls
Brief Title: Pharmacokinetics of Vitamin D in Multiple Sclerosis and in Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: University of California, San Francisco (Other); National Multiple Sclerosis Society (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NA_00049428; FG-1507-05231 (Other Grant/Funding Number: National Multiple Sclerosis Society)
Record Dates: First submitted 2012-08-13; First posted 2012-08-17 (Estimated); Results first posted 2016-02-01 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Multiple Sclerosis, Relapsing-remitting
Keywords: Multiple sclerosis; Healthy controls; Pharmacokinetics; Vitamin D
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vitamin D3 (Experimental): Both those with MS and healthy controls will be given vitamin D3 5000 IU/day by mouth for 90 days.
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D3

SUMMARY:
This is a pilot study of oral vitamin D supplementation to determine if patients with Multiple Sclerosis (MS) and healthy individuals attain a similar increase in serum 25-hydroxyvitamin D levels. The investigators will also assess whether the immunologic or relevant gene expression response to oral vitamin D supplementation differs in patients with MS and healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Healthy or multiple sclerosis
* Aged 18 to 60
* Body mass index is between 18 kg/m2 and 30 kg/m2
* Screening 25-hydroxyvitamin D level ≤ 75 nmol/L (30 ng/mL)
* White race
* Non-Hispanic ethnicity
* Willing to use birth control during study
* Willing to not use tanning bed during study

If subject has multiple sclerosis:

* Relapsing-remitting MS, as defined by McDonald 2005 criteria
* Screening Expanded Disability Status Scale score ≤ 3.0
* Using no medication for MS, or taking Copaxone, (glatiramer acetate), interferons, or natalizumab

Exclusion Criteria:

* Pregnant or nursing
* Taking multivitamin & unwilling to remain off it during study
* Taking cod liver oil & unwilling to remain off it during study
* On a fat-restricted diet
* History of renal disease or nephrolithiasis (kidney stones)
* History of liver disease
* Taking thiazide diuretics
* History of hyperthyroidism
* History of infection with Mycobacterium species
* History of sarcoidosis
* History of cancer
* History of cardiac disease
* History of HIV
* History of gastrointestinal disorder
* Taking medications that interfere with gastrointestinal absorption
* Cigarette smoker in past month
* Use of illicit drugs in past month
* Use of steroids in past month
* History of hypercalcemia, and screening serum calcium ≤ 10 mg/dL (UCSF) or ≤ 10.7 mg/dL (Johns Hopkins)
* History of hypercalciuria
* Evidence of anemia (Hgb <11.0 g/dL)
* History of other serious medical conditions
* Taking medications that involve the P450 system or may interact with vitamin D (digoxin, diltiazem, verapamil, cimetidine, heparin, or low-molecular weight heparin)
* Other concerns about safety from the perspective of the treating physician

If subject has MS:

-History of major heat sensitivity (leading to sun-avoidant behaviors)

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2010-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen M Mowry, MD, MCR, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - Johns Hopkins University, Baltimore, Maryland

REFERENCES:
- [Derived] Bhargava P, Fitzgerald KC, Calabresi PA, Mowry EM. Metabolic alterations in multiple sclerosis and the impact of vitamin D supplementation. JCI Insight. 2017 Oct 5;2(19):e95302. doi: 10.1172/jci.insight.95302. PMID 28978801

RESULTS

PARTICIPANT FLOW:
Groups:
- Multiple Sclerosis (MS) Subjects: MS patients
- Healthy Controls: Healthy control subjects
Period: Overall Study
Arm/Group | Multiple Sclerosis (MS) Subjects | Healthy Controls
Started | 27 | 30
Completed | 24 | 29
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- MS Subjects: Female subjects with MS
- Healthy Controls: Female subjects without MS
- Total: Total of all reporting groups
Arm/Group | MS Subjects | Healthy Controls | Total
Number analyzed (Participants) | 27 | 30 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.2 (9.2) | 37.9 (12.1) | 38.9 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 30 | 57
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 27 | 30 | 57
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 27 | 30 | 57

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Serum Level of 25-hydroxyvitamin D
Description: Generalized estimating equations (GEE) with an autoregressive with lag one correlation matrix were used to compare the serially-measured serum 25(OH)D levels between MS patients and Healthy Controls (HCs) to take into account repeated measures and within-subject correlations.
Time Frame: Baseline to 90 days
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | MS Subjects | Healthy Controls
Number analyzed (Participants) | 24 | 29
nmol/L | 65.9 (5.9) | 82.4 (5.2)
Statistical Analysis 1: Comparison: MS Subjects vs Healthy Controls; Test type: Superiority or Other; p = 0.001, univariate generalized estimating equati
Statistical Analysis 2: Comparison: MS Subjects vs Healthy Controls; Test type: Superiority or Other; p = 0.008, Generalized estimating equation — Adjusted for adherence, body mass index, and oral contraceptive use

2. Secondary Outcome: Change in Percentages of T Cell Subsets (IFNγ+ and IL-17+)
Description: Analyzed the mean percentage change in IFNγ+ and IL-17+ cluster of differentiation 4 (CD4) + cells (post- versus pre- supplementation). This represents a change between two time points (90 days versus baseline).
Time Frame: Baseline, 90 days
Measure: Mean (Standard Deviation); unit: percentage of cells
Groups:
- MS Subjects: MS patients
Arm/Group | MS Subjects | Healthy Controls
Number analyzed (Participants) | 11 | 14
percentage of cells
  mean percentage change in IFNγ+ CD4+ cells | -5.2 (4.2) | -13.2 (3.2)
  mean percentage change in IL-17+ CD4+ cells | 0.21 (0.77) | -0.17 (1.14)

3. Secondary Outcome: Gene Expression Microarray
Description: We had initially planned to do whole blood gene expression. The experience gained by the laboratory that was to perform this since the original trial was planned was that this measure is too noisy and would not yield meaningful results. Thus, this analysis will no longer be conducted.
Time Frame: 90 days
Population: We had initially planned to do whole blood gene expression. The experience gained by the laboratory that was to perform this since the original trial was planned was that this measure is too noisy and would not yield meaningful results. Thus, this analysis will no longer be conducted.
Groups:
- Gene Expression: MS vs HC: Gene expression analyses have been cancelled as a secondary outcome as laboratory techniques developed since the original study was started indicated that whole blood gene expression is unlikely to be informative.
Arm/Group | Gene Expression: MS vs HC
Number analyzed (Participants) | 0

4. Secondary Outcome: Change in Cytokine Levels
Description: The original plan had been to measure the change in basic serum cytokine levels (e.g. IL-17, interferon gamma; IL-10; pg/microliter). However, due to emerging data suggesting low utility of these measures, this plan was abandoned.
Time Frame: 90 days
Population: Cytokine levels data were not analyzed and are no longer planned to be measured as outcomes.
Arm/Group | Multiple Sclerosis (MS) Subjects | Healthy Controls
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Percentage of B Cells
Description: The change in percentage (day 90-baseline) was originally planned for study. Due to the limited number of patients with samples this plan was abandoned.
Time Frame: 90 days
Population: B Cell data were not analyzed and are no longer planned to be measured as outcomes.
Arm/Group | Multiple Sclerosis (MS) Subjects | Healthy Controls
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | MS Subjects | Healthy Controls
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/30
Other Adverse Events (participants affected / at risk) | 0/27 | 1/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MS Subjects (N=27) | Healthy Controls (N=30)
Palpitations (Cardiac disorders) | 0 | 1 — A control got palpitations. Cardiac workup: rare premature atrial and ventricular contractions; the person then reported remote atrial fibrillation (not disclosed at screening visit). This was not deemed to be related to vitamin D supplementation.

LIMITATIONS AND CAVEATS:
The generalizability of the findings of this study (beyond female Caucasians) has to be further tested. It is possible that there were unmeasured confounders influencing results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No